CLINICAL TRIAL: NCT00004996
Title: Langherhans' Cell Function and Inflammatory Responses in Skin of Volunteers Using the Suction Blister Technique
Brief Title: Comparison of Immune Response in Normal Volunteers and Patients With Helminth Infections
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000099; 00-I-0099
Record Dates: First submitted 2000-03-22; First posted 2000-03-23 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2015-04-22

CONDITIONS: Healthy; Helminthiasis
Keywords: Antigen Presentation; Cytokines; Helminth; Healthy Volunteer; Cross-Over Study; Helminth Infection
MeSH Terms: conditions — Helminthiasis; Trematode Infections

SUMMARY:
This study will compare the structure, chemical composition and other characteristics of skin and blood in people with and without parasitic infections. Cell samples will be taken from blisters produced by suction blistering. This study may provide new information about the interactions between parasites and the immune system that could lead to better treatments for these infections.

Normal volunteers and patients with acute helminth (a type of parasite) infections aged 18 years older may be eligible for this study. Following a medical history and physical exam, participants will undergo suction blistering to provide cells needed for study. A suction blister device is attached to the skin of the thigh. A heating element in the device heats the skin to speed blister formation. (This will feel only a slightly warm.) The device is removed after about two hours, when the blisters have formed. The blister tops are removed with sterile scissors. The blistered areas are then treated with special dressings to promote healing and the participant is discharged with further wound care instructions. A small amount of blood (around four tablespoons) may be drawn to compare chemicals in the blood with chemicals in the blister fluid. Participants will be contacted by telephone over the next 72 hours to check on healing. Further follow-up will occur by phone at 6 months and 1 year.

Up to 60 blisters may be produced over a one-year period (in three separate sessions every six months) with no more than 20 raised per session....

DETAILED DESCRIPTION:
This study will compare the structure, chemical composition and other characteristics of skin and blood in people with and without parasitic infections. Cell samples will be taken from blisters produced by suction blistering. This study may provide new information about the interactions between parasites and the immune system that could lead to better treatments for these infections.

Normal volunteers and patients with acute helminth (a type of parasite) infections aged 18 years older may be eligible for this study. Following a medical history and physical exam, participants will undergo suction blistering to provide cells needed for study. A suction blister device is attached to the skin of the thigh. A heating element in the device heats the skin to speed blister formation. (This will feel only a slightly warm.) The device is removed after about two hours, when the blisters have formed. The blister tops are removed with sterile scissors. The blistered areas are then treated with special dressings to promote healing and the participant is discharged with further wound care instructions. A small amount of blood (around four tablespoons) may be drawn to compare chemicals in the blood with chemicals in the blister fluid. Participants will be contacted by telephone over the next 72 hours to check on healing. Further follow-up will occur by phone at 6 months and 1 year.

Up to 60 blisters may be produced over a one-year period (in three separate sessions every six months) with no more than 20 raised per session.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Between the ages of 18 and 65 years inclusive
  2. Access to a primary medical care provider outside of the NIH
  3. Able to give informed consent
  4. Willingness to have history and physical examination annually

EXCLUSION CRITERIA:

1. History of malignancy or autoimmune disease such as rheumatoid arthritis, vasculitis, pyoderma gangrenosum
2. Use of systemic corticosteroids within the past month
3. Use of local corticosteroids at the proposed blistering site within the past month
4. Evidence of current acute infection
5. Personal or family history of keloid formation
6. Use of any investigative drugs within the past month
7. History of skin disease within the past one year (e.g. psoriasis, atopic dermatitis)
8. History of diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2000-03-20; Study Completion 2015-04-22

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B Nutman, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kiistala U. Suction blister device for separation of viable epidermis from dermis. J Invest Dermatol. 1968 Feb;50(2):129-37. doi: 10.1038/jid.1968.15. No abstract available. PMID 4868034
- [Background] Blauvelt A, Katz SI, Udey MC. Human Langerhans cells express E-cadherin. J Invest Dermatol. 1995 Feb;104(2):293-6. doi: 10.1111/1523-1747.ep12612830. PMID 7829887
- [Background] Dale DC, Wolff SM. Skin window studies of the acute inflammatory responses of neutropenic patients. Blood. 1971 Aug;38(2):138-42. No abstract available. PMID 4933314